CLINICAL TRIAL: NCT03600571
Title: Injection Site Diversity Influences Sodium Hyaluronate Distribution and Its Clinical Results in Management of Chondromalacia Patellae and Knee Osteoarthritis: A Preliminary, Multi-central, Randomize-controlled Serial Trial
Brief Title: Injection Site Diversity Influences HA Distribution and Clinical Results in CP and KOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2014-074
Record Dates: First submitted 2018-06-30; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis, Knee; Hyaluronan
Keywords: Viscosupplementation; Hyaluronate; Distribution; Knee osteoarthritis; Injection approach
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Matrix Metalloproteinases

STUDY DESIGN:
Intervention Model Description: 64 osteoarthritic knees of cadavers were randomly assigned to two groups: the anteromedial (AM) group (n=32) and the medial midpatellar (MMP) group (n=32).
  100 patients with unilateral mKOA were enrolled and randomly divided into two groups according to the injection portal of HA: the AM group (n=50) and the MMP group (n=50).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AM groups in cadavers study (Experimental): 32 osteoarthritic knees of cadavers were randomly assigned to the AM group (injection medial from patella tendon towards intercondylar notch was performed with the target knee 90° flexion). Hyaluronic acid (HA) traced by methylene blue was injected into the knee, and the intra-articular distribution of HA was assessed using a five-point scale.
  Interventions: Procedure: anteromedial (AM) portal
- MMP groups in cadavers study (Experimental): 32 osteoarthritic knees of cadavers were randomly assigned to the MMP group (injection medial under horizontal patella midline was administrated with the lower limb extension). Hyaluronic acid (HA) traced by methylene blue was injected into the knee, and the intra-articular distribution of HA was assessed using a five-point scale.
  Interventions: Procedure: medial midpatellar (MMP) portal
- AM groups in random controlled trial (Experimental): 50 patients with unilateral mKOA were enrolled and randomly into the AM group (injection medial from patella tendon towards intercondylar notch was performed with the target knee 90° flexion).The clinical outcomes of 5-weekly injections of HA were evaluated by WOMAC and Lequesne index. The follow-up times were at weeks 1, 2, 3, 4, 5, 14, and 24 after the injections.
  Interventions: Procedure: anteromedial (AM) portal
- MMP groups in random controlled trial (Experimental): 50 patients with unilateral mKOA were enrolled and randomly into the MMP group (injection medial under horizontal patella midline was administrated with the lower limb extension).The clinical outcomes of 5-weekly injections of HA were evaluated by WOMAC and Lequesne index. The follow-up times were at weeks 1, 2, 3, 4, 5, 14, and 24 after the injections.
  Interventions: Procedure: medial midpatellar (MMP) portal

INTERVENTIONS:
Procedure: medial midpatellar (MMP) portal — injection medial under horizontal patella midline was administrated with the lower limb extension
  Arms: MMP groups in cadavers study; MMP groups in random controlled trial
Procedure: anteromedial (AM) portal — injection medial from patella tendon towards intercondylar notch was performed with the target knee 90° flexion
  Arms: AM groups in cadavers study; AM groups in random controlled trial

SUMMARY:
In order to investigate the difference of intra-articular hyaluronate's distribution and compare the clinical outcomes of viscosupplementation for mild-to-moderate knee osteoarthritis (mKOA) between the anteromedial (AM) and medial midpatellar (MMP) approach groups. This study included two parts, cadaver study (n=64) and random controlled trial (n=100). Hyaluronic acid (HA) traced by methylene blue was injected into the knee, and the intra-articular distribution of HA was assessed using a five-point scale in the cadaver study. The clinical outcomes of 5-weekly injections of HA were evaluated by WOMAC and Lequesne index and the follow-up times were at weeks 1, 2, 3, 4, 5, 14, and 24 after the injections in the random controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic unilateral mild-to-moderate knee osteoarthritis (mKOA) that were defined by the American College of Rheumatology criteria
* Kellgren-Lawrence grade 2 or 3
* Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index (Likert version 3.1) pain subscale reached 10 or greater

Exclusion Criteria:

* Pregnancy, acute fracture, rheumatoid arthritis, gouty arthritis, traumatic arthritis, inflammatory arthritis
* Oral Celebrex within 2 weeks, HA and lidocaine allergy, intra-articular injection of HA or corticosteroid to the target knee within the past 6 months
* Surgery in the target knee within the past 6 months, OA of the target knee with K-L grade 4
* Active liver and renal disease, cardiovascular and cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-08-30 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
WOMAC (Likert version 3.1) | baseline before the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 1 week after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 2 weeks after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 3 weeks after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 4 weeks after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 5 weeks after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 14 weeks after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
WOMAC (Likert version 3.1) | 24 weeks after the first injection
  WOMAC included three subscales: pain, stiffness and function, and each subscale was graded using a 5-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Pain index score ranges from 0 to 20, whereas the stiffness score ranges from 0 to 8 and the function score ranges from 0 to 68. The reliability of the three subscales of the WOMAC was 0.82, 0.68 and 0.74, respectively.
Lequesne index | baseline before the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 1 week after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 2 weeks after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 3 weeks after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 4 weeks after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 5 weeks after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 14 weeks after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.
Lequesne index | 24 weeks after the first injection
  The Lequesne index questionnaire included 10 questions about pain, stiffness and function. The score ranges from 0 (no pain, no disability) to 24 (maximum pain, stiffness and disability), and its reliability was 0.95.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China